CLINICAL TRIAL: NCT00091871
Title: A Longitudinal Study of Familial Hypereosinophilia (FE): Natural History and Markers of Disease Progression
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040286; 04-I-0286
Record Dates: First submitted 2004-09-17; First posted 2004-09-20 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-05-15

CONDITIONS: Eosinophilia; Hypereosinophilic Syndrome
Keywords: Hypereosinophilia; Eosinophil; Familial; Interleukin 5; Natural History; Familial Hypereosinophilia; FE
MeSH Terms: conditions — Eosinophilia; Hypereosinophilic Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected family members: Family members with peripheral blood eosinophilia
- Unaffected family members: Family members without peripheral blood eosinophilia

SUMMARY:
Eosinophils are a type of white blood cell. Elevated eosinophil levels can damage the heart, nerves, and other organs, in the syndrome known as hypereosinophilic syndrome (HES). Some individuals have a hereditary form of HES known as familial eosinophilia (FE). More research on the causation and mechanisms of HES is needed in order to design more effective and less toxic therapies.

This study will investigate FE and its genetic causes, damage mechanisms, and disease markers (such as blood test abnormalities). It will enroll approximately 50 individuals (both adults and children) from a previously studied family with FE. This is a long-term study of indefinite duration.

Participants will undergo yearly clinical examinations including medical history, physical examination, bloodwork, EKG, echocardiogram, and pulmonary function tests, with additional or more frequent examinations and tests as required. In addition, participants will donate blood and tissue for research purposes. Both adult and child participants will donate blood. At the initial evaluation, adult participants will donate bone marrow. During the study, some adult participants will also undergo a limited number of leukaopheresis sessions, in which blood is donated from one arm, the blood is separated into red blood cells and other components, and the red blood cells are returned into the donor's other arm.

DETAILED DESCRIPTION:
Study Description:

Affected and unaffected members of families with familial hypereosinophilia (FE) will be enrolled and evaluated on this protocol. For affected family members, a thorough clinical evaluation will be performed with emphasis on potential sequelae of eosinophil-mediated tissue damage. Blood cells, bone marrow and/or serum will also be collected to provide reagents (such as DNA, RNA, and specific antibodies) for use in the laboratory to address issues related to the genetic and immunologic basis of FE as well as its pathogenesis. It is anticipated that affected family members will undergo a more extensive evaluation than is generally available and that the specimens collected from them will prove to be valuable reagents for laboratory studies related to eosinophilia, eosinophil activation and function. While the study is not designed to address the question of therapy for FE, in patients for whom medical therapy is indicated (for either the hypereosinophilia itself or its sequelae), appropriate treatment will be instituted by our clinical service or the patients local physicians. No experimental chemotherapy is involved in this protocol. Unaffected family members will provide research specimens on this protocol to help determine the underlying genetic causes of FE.

Objectives:

Primary Objective: To study the natural history of familial hypereosinophilia (FE)

Secondary Objectives:

1. To determine the immunologic and molecular mechanisms responsible for eosinophilia, eosinophil activation, and pathogenesis in FE
2. To identify early clinical or laboratory markers of disease progression

Endpoints: Primary Endpoint: Development of eosinophilic end organ manifestations

Secondary Endpoints:

1a. Description of immunologic features of FE.

1b. Identification of genetic driver(s) of FE

2. Identification of clinical or laboratory markers that become abnormal prior to disease progression in FE

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 1-100 years of age
* Genetically related member of a previously identified family with FE
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any condition that the investigator feels put the subject at unacceptable risk for participation in the study
* Pregnancy (in family members who do not have eosinophilia)

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Affected family members from the previously identified family with FE, as well as affected member of newly identified families with FE and unaffected family members from known families with FE, may enroll.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-06-08 (Actual)

PRIMARY OUTCOMES:
To study the natural history of familial hypereosinophilia (FE) | 30 years
  Development of eosinophilic end organ manifestations

SECONDARY OUTCOMES:
To determine the immunologic and molecular mechanisms responsible for eosinophilia, eosinophil activation, and pathogenesis of FE | 30 years
  Description of immunologic features of FE; identification of genetic driver(s) of FE
To identify early clinical or laboratory markers of disease progression | 30 year
  Identification of clinical or laboratory markers that become abnormal prior to disease progression in FE

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a longitudinal observational study in a rare inherited disease. At this point in time, there is no plan to share individual participant data as the main outcomes of the study are based on group data (incidence of end organ manifestations in the group) and identification of genetic and immunologic drivers of familial eosinophilia.

REFERENCES:
- [Background] Rioux JD, Stone VA, Daly MJ, Cargill M, Green T, Nguyen H, Nutman T, Zimmerman PA, Tucker MA, Hudson T, Goldstein AM, Lander E, Lin AY. Familial eosinophilia maps to the cytokine gene cluster on human chromosomal region 5q31-q33. Am J Hum Genet. 1998 Oct;63(4):1086-94. doi: 10.1086/302053. PMID 9758611
- [Background] Prakash Babu S, Chen YK, Bonne-Annee S, Yang J, Maric I, Myers TG, Nutman TB, Klion AD. Dysregulation of interleukin 5 expression in familial eosinophilia. Allergy. 2017 Sep;72(9):1338-1345. doi: 10.1111/all.13146. Epub 2017 Apr 18. PMID 28226398
- [Background] Klion AD, Law MA, Riemenschneider W, McMaster ML, Brown MR, Horne M, Karp B, Robinson M, Sachdev V, Tucker E, Turner M, Nutman TB. Familial eosinophilia: a benign disorder? Blood. 2004 Jun 1;103(11):4050-5. doi: 10.1182/blood-2003-11-3850. Epub 2004 Feb 26. PMID 14988154
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-I-0286.html